CLINICAL TRIAL: NCT01245361
Title: "A Comparative Study Of A 6-Month Infliximab (Remicade®) Or Placebo Regimen In Undifferentiated Arthritis At High Risk For The Development Of Rheumatoid Arthritis (RA) : Clinical, Radiological (MRI) And Synovial Benefit P1200/001".
Brief Title: A 6-Months Infliximab Or Placebo Study In UA At High Risk Of RA:Clinical,Radiological And Synovial Benefit
Acronym: UA-IFX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Durez (Other)
Responsible Party: Sponsor-Investigator, Patrick Durez, Professor, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P1200/001
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Undifferentiated Arthritis
Keywords: Undifferentiated Arthritis; Rheumatoid Arthritis; Infliximab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab (Experimental): Group I: Infliximab 3 mg/kg wk 0,2,6
  Interventions: Drug: Infliximab
- sodium chloride (Placebo Comparator): RA 1 solution for infusion, intravenous use Sterile normal saline 0.9% sodium chloride
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: Infliximab — Infliximab 3 mg/kg wk 0,2,6
  Other Names: FR-BR7794
  Arms: Infliximab
Drug: sodium chloride — Group II : Placebo wk 0,2,6
  Arms: sodium chloride

SUMMARY:
Patient with undifferentiated arthritis and the presence of anti-citruline (anti-CCP) antibodies are at high risk to develop RA. The presence of anti-CCP is associated with a higher rate of erosion and a higher risk of progressive and severe RA.

The investigators have demonstrated in the CIERA study that MTX/IFX combination therapy is superior to MTX alone to reduce MRI signs of synovitis and bone edema and is clinically more effective.

The immunopathogenesis of undifferentiated arthritis is poorly understood. However, synovial studies from patients with early arthritis suggest that UA and RA may share common immunopathogenic mechanisms. One biopsy study of asymptomatic joints in patients with early arthritis demonstrates synovitis in more than half of the joints samples with prominent T cell and macrophage infiltration, similar to Rheumatoid Arthritis (RA).

Thus intensive treatment with anti-TNF antibodies (infliximab) may have an impact on multiple immune mechanisms driving synovitis in undifferentiated arthritis and may influence the clinical outcome.

Recently, Methotrexate has been demonstrated to improve the course of undifferentiated arthritis and prevent the development of RA. Short regimen of more intensive therapy with Infliximab could alter the radiological, immunopathological and clinical outcome.

DETAILED DESCRIPTION:
not necessary

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of UA Absence of American College of Rheumatology (ACR) criteria Active UA defined by a swollen joint count ≥ 1 and < 4 Positive anti-CCP Disease duration < 2 years DMARDs naive No chronic treatment with steroids (> 3 months), if needed washout of 4 weeks NSAIDs stable

Exclusion Criteria:

Other rheumatic inflammatory diagnosis Contraindication to MRI (pace-maker, etc.) Congestive heart disease Active or latent tuberculosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary objective To compare the induction therapy with infliximab versus placebo on the MRI synovitis and erosion score in undifferentiated arthritis. | 2 years
  not necessary

SECONDARY OUTCOMES:
To test the hypothesis that induction therapy with infliximab is followed by a better clinical outcome over a 2 year follow-up and defined as a lower rate of patients with ACR criteria at 6, 12 and 24 months. | 2 years
  no necessary
To assess the effects of infliximab on synovial histopathology of UA. | 2 years
  no necessary
To test the hypothesis that infliximab can influence the presence of anti CCP antibodies. | 2 years
  no necessary
To assess physical function and health-related quality of life using the Disability Index of HAQ (HAQ) and questionnaire "SF-36" instruments, respectively | 2 years
  no necessary

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Durez, Md, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain, Brussels, Belgium